CLINICAL TRIAL: NCT04712695
Title: Comparing the Effectiveness of Various Interventions on Improving Lumbar Proprioception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Black Hills State University (Other)
Responsible Party: Principal Investigator, Craig Triplett, Associate Professor Exercise Science, Black Hills State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BlackHillsSU
Record Dates: First submitted 2021-01-12; First posted 2021-01-15 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Proprioception

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Graded Motor Imagery Group (Experimental)
  Interventions: Other: Exercise Based Interventions
- Mirror Visual Feedback Group (Experimental)
  Interventions: Other: Exercise Based Interventions
- Augmented Biofeedback Group (Experimental)
  Interventions: Other: Exercise Based Interventions
- Diaphragmatic Breathing Group (Sham Comparator)
  Interventions: Other: Exercise Based Interventions

INTERVENTIONS:
Other: Exercise Based Interventions — Proprioception Training Interventions

SUMMARY:
University students ages 18-45, with no recent history of back injury and no history of back surgery, were recruited. Participants completed proprioception testing consisting of a standing side bending and seated spinal flexion test. Participants performed each test once, then were blindfolded and asked to replicate the tests 10 times. After the initial proprioceptive testing, the participants were randomly split into four groups and performed a 10-minute intervention exercise, before repeating the proprioceptive tests for final measurements. The four groups included: graded motor imagery, mirror visual feedback, augmented biofeedback, and diaphragmatic breathing. Participants also completed a Physical Activity Enjoyment Scale to rate their enjoyment of their intervention task

-For the seated forward flexion test, the participants' C7 and S2 vertebrae were identified and used as markers. The participants were asked to bend forward until the tape measure increased 5 cm from the original distance between the C7 and S2 vertebrae. Similar to the seated flexion test, during the side-bending task, the participants were asked to side bend until the tip of their middle finger was 10 cm closer to the floor. The participants were asked to memorize that point in their mind; they were then blindfolded and asked to repeat the movement 10 times, trying to recreate the original position to the best of their ability.

Between initial and final measurements of proprioception, the participants were randomly assigned to one of the following four groups for interventions for a 10-minute training session:

* Graded Motor Imagery Group: Participants were shown several flashcards with pictures of individuals' back oriented to either the flexed or side bent position. The participants stated which direction the image depicted and visualized themselves making the movement identified in the picture.
* Mirror Visual Feedback Group:

Participants viewed themselves in a mirror while performing flexion and side bending movements.

-Augmented Biofeedback Group: Participants used an augmented musculoskeletal feedback system smartphone application app and small sensors with Bluetooth technology to translate the movement of the participant into an avatar on the game.

-Diaphragmatic Breathing Group: Participants were told to sit on a chair with their back straight and feet flat on the floor with one hand on their chest and one hand on their stomach. They performed diaphragmatic breathing in a slow 4 second box method: breathing in for 4 seconds, holding for 4 seconds, breathing out for 4 seconds, and then hold for 4 seconds

ELIGIBILITY:
Inclusion Criteria:

* Healthy university students ages 18-35
* Must be able to perform low intensity exercise

Exclusion Criteria:

* Past medical history of back surgery
* Back pain within the past 6 months
* Musculoskeletal injury within the past 6 months

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Proprioception | Day 1
  Change in lumbar proprioception as assessed through the seated forward flexion test measured in cm following a single training session.

CONTACTS AND LOCATIONS:
Locations (1):
- Black Hills State University, Spearfish, South Dakota, United States

IPD SHARING:
Plan to Share IPD: Undecided